CLINICAL TRIAL: NCT01402141
Title: Efficacy and Safety of Chungkookjang, a Fermented Soy Paste, on Histamine-induced Wheal Size
Brief Title: A Human Trial to Evaluate the Effects of Chungkookjang on Histamine-induced Wheal Size in Healthy Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SunChang-TCKJ-001
Record Dates: First submitted 2011-07-21; First posted 2011-07-26 (Estimated); Results first posted 2012-11-12 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Healthy Subjects
Keywords: Chungkookjang; histamine; skin reaction; wheal
MeSH Terms: conditions — Urticaria | interventions — chungkookjang

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chungkookjang (Experimental)
  Interventions: Dietary Supplement: Chungkookjang
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Chungkookjang — Chungkookjang(35g/say)for 12 weeks
  Arms: Chungkookjang
Dietary Supplement: Placebo — Placebo(35g/day) for 12 weeks
  Arms: Placebo

SUMMARY:
The investigators investigate the effect of Chungkookjang on histamine-induced skin reaction in a double-blind, randomized, placebo-controlled, human trial

DETAILED DESCRIPTION:
Sixty volunteers (aged 20-80) who gave a written consent before entering the study, were randomized in two groups of thirty subjects each. The skin prick test with histamine was performed on the ventral forearm, 10 cm from the elbow, before and after supplement administration, as well as three times daily for 12 weeks of chungkookjang(35g/day) or placebo(35g/day)intake.

ELIGIBILITY:
Inclusion Criteria:

* Histamine skin prick test: above 3mm

Exclusion Criteria:

* No medication or cosmetic creams were allowed during Substances the previous week and no drugs containing corticosteroids or ACTH within 3 months.
* Patients on systemic or topical treatment with immunosuppressive agents on the nondominant arm were excluded

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baek-Hwan Cho, MD., PhD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

REFERENCES:
- [Derived] Kwon DY, Yang HJ, Kim MJ, Kang HJ, Kim HJ, Ha KC, Back HI, Kim SY, Park EO, Kim MG, Yun SK, Chae SW, Cho BH. Influence of the Chungkookjang on histamine-induced wheal and flare skin response: a randomized, double-blind, placebo controlled trial. BMC Complement Altern Med. 2011 Dec 5;11:125. doi: 10.1186/1472-6882-11-125. PMID 22136279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through local advertising and doctor referrals from hospital outpatients and general practice clinics.
Pre-assignment Details: The criteria were an age from 19 to 80 years, Histamine skin prick test: above 3mm
Groups:
- Chungkookjang: Chungkookjang(3times/day, 3packs/day, 35g/day) for 12weeks
  Chungkookjang: The Chungkookjang was manufactured from raw beans, peels made after freeze-drying
- Placebo: Placebo(3times/day, 3packs/day, 35g/day) for 12weeks
  Placebo : Amount and calorie of placebo are same with Chungkookjang.
Period: Overall Study
Arm/Group | Chungkookjang | Placebo
Started | 30 | 30
Completed | 29 | 28
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chungkookjang(35g) | Placebo(35g) | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.5 (11.9) | 34.2 (12.9) | 34.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 28 | 48
  Male | 10 | 2 | 12
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Changes in Histamine-induced Wheal Size
Description: Histamine-induced wheal size was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: mm^2
Groups:
- Chungkookjang: Oral intake Chungkookjang(35g) for 12weeks.
- Placebo: Oral intake placebo(35g/day) for 12weeks
Arm/Group | Chungkookjang | Placebo
Number analyzed (Participants) | 29 | 28
mm^2
  Pre | 14.9 (7.3) | 14.9 (7.0)
  Post | 14.1 (7.7) | 16.5 (5.8)

2. Secondary Outcome: Changes in Immunoglobulin E
Description: Immunoglobulin E was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Chungkookjang | Placebo
Number analyzed (Participants) | 29 | 28
IU/mL
  Pre | 73.89 (92.38) | 69.32 (110.25)
  Post | 67.32 (81.74) | 62.72 (96.53)

3. Secondary Outcome: Changes in Serum Histamine
Description: Serum histamine was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: μg/g creatinine
Arm/Group | Chungkookjang | Placebo
Number analyzed (Participants) | 29 | 28
μg/g creatinine
  Pre | 0.56 (0.54) | 0.62 (0.51)
  Post | 0.79 (0.58) | 0.80 (0.73)

4. Secondary Outcome: Changes in Interferon-gamma
Description: Interferon-gamma was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: IU/ml
Arm/Group | Chungkookjang | Placebo
Number analyzed (Participants) | 29 | 28
IU/ml
  Pre | 14.56 (3.08) | 15.63 (5.46)
  Post | 17.57 (1.87) | 18.06 (2.22)

5. Secondary Outcome: Changes in Interleukin-4
Description: Interleukin-4 was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Chungkookjang | Placebo
Number analyzed (Participants) | 29 | 28
pg/ml
  Pre | 0.78 (0.78) | 0.55 (1.56)
  Post | 0.26 (0.20) | 0.35 (0.78)

6. Secondary Outcome: Changes in Eosinophil
Description: Eosinophil was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: Percentage of WBCs(white blood cells)
Arm/Group | Chungkookjang | Placebo
Number analyzed (Participants) | 29 | 28
Percentage of WBCs(white blood cells)
  Pre | 2.66 (2.14) | 3.30 (2.87)
  Post | 2.54 (2.23) | 2.56 (2.56)

7. Secondary Outcome: Changes in Eosinophil Cationic Protein(ECP)
Description: Eosinophil Cationic Protein(ECP) was measured in study visit 1(0 week) and visit 3(12 week).
Time Frame: 12weeks
Population: per protocol analysis
Measure: Mean (Standard Deviation); unit: μg/L
Groups:
- Placeb: Oral intake placebo(35g/day) for 12weeks
Arm/Group | Chungkookjang | Placeb
Number analyzed (Participants) | 29 | 28
μg/L
  Pre | 17.55 (17.28) | 23.53 (21.00)
  Post | 19.09 (17.49) | 21.80 (26.10)

8. Primary Outcome: Number of Participants With Greater Than 40% Decrease in Histamine-induced Wheal Size (Wheal Size by More Than 40% Decrease in the Number of Subjects Compared With Placebo)
Description: Number of Participants with Greater than 40% Decrease in Histamine-induced Wheal Size was measured in study visit 1(0 week) and visit 3(12 week).
  Percentage change in histamine-induced wheal size calculations were calculated by the formula ((12weeks - 0weeks) * 100/0weeks).
  Number of Participants with Greater than 40% Decrease in Histamine-induced Wheal Size compared with placebo.
Time Frame: 12weeks
Population: per protocol analysis
Measure: Number; unit: participants
Arm/Group | Chungkookjang | Placebo
Number analyzed (Participants) | 29 | 28
participants | 6 | 1

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Groups:
- Chungkookjang(35g): Oral intake Chungkookjang(35g) for 12weeks.
- Placebo(35g): Oral intake placebo(35g/day) for 12weeks
Arm/Group | Chungkookjang(35g) | Placebo(35g)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No